CLINICAL TRIAL: NCT07078344
Title: Addressing Diet-Induced Health Disparities With Precision Nutrition and Omega-3 Fatty Acids
Brief Title: Omega-3D: Omega-3 for Diet-Driven Health Disparities
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Arizona (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Georgetown University (Other)
Responsible Party: Principal Investigator, Patricia Thompson, Professor of Physiology, University of Arizona
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: STUDY00005456; 2R01AT008621-07 (NIH)
Record Dates: First submitted 2025-04-10; First posted 2025-07-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Heart Health Markers; Cardiovascular Diseases; Omega 3 Fatty Acids
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identical capsules and packaging for omega-3 and safflower oil placebo; blinded allocation and crossover order.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blinded Crossover Arm: Omega-3 Fatty Acids and Safflower Oil Placebo (Experimental): Participants receive both study interventions (omega-3 fatty acid supplement and safflower oil placebo) across two blinded treatment periods in a randomized crossover design. The randomization schedule determines which supplement is administered first, but participants and investigators remain blinded to the identity and order of study supplements.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids and Safflower Oil Placebo; Dietary Supplement: Safflower Oil Placebo and Omega-3 Fatty Acids
- Blinded Crossover Arm: Safflower Oil Placebo and Omega-3 Fatty Acids (Experimental): Participants receive both study interventions (safflower oil placebo and omega-3 fatty acid supplement) across two blinded treatment periods in a randomized crossover design. The sequence is the opposite of Arm 1, but study blinding prevents participants and investigators from knowing which supplement is administered during each period.
  Interventions: Dietary Supplement: Omega-3 Fatty Acids and Safflower Oil Placebo; Dietary Supplement: Safflower Oil Placebo and Omega-3 Fatty Acids

INTERVENTIONS:
Dietary Supplement: Omega-3 Fatty Acids and Safflower Oil Placebo — Blinded study supplement; appearance-matched softgels.
Dietary Supplement: Safflower Oil Placebo and Omega-3 Fatty Acids — Blinded study supplement; appearance-matched softgels.

SUMMARY:
The goal of this clinical trial is to learn whether omega-3 fatty acid supplementation can reduce inflammation-related biomarkers and improve cardiovascular health in healthy adult volunteers with different genetic backgrounds. The main questions it aims to answer are: Does the response to omega-3 supplementation differ based on genetic variation in the FADS gene cluster (specifically rs174537)? Are changes in fatty acid ratios and inflammation markers greater among individuals of African ancestry compared to those of European ancestry? Researchers will compare omega-3 supplements to a placebo in a randomized, placebo-controlled crossover study to determine whether the Omega-3 supplementation is more effective in certain genetic and ancestry groups. Participants will take omega-3 supplements or a placebo daily for a defined period, then cross over to the other intervention. They will provide blood samples for analysis of fatty acid levels and inflammatory markers, complete questionnaires, and attend scheduled study visits.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≥ 18.5 kg/m2
* Self-identify as non-Hispanic African American or non-Hispanic European American
* Ability and willingness to transport for regular clinic visits.
* Ability and willingness to swallow study capsules.
* Willingness to refrain from intentional weight loss
* Willingness maintain usual physical activity levels and dietary intake throughout the trial.

Exclusion Criteria:

* Age > 65 years
* BMI ≥ 40 kg/m2
* Currently pregnant or breastfeeding.
* Currently receiving treatment for cancer (excluding adjuvant therapies).
* Consumption of DHA/EPA-rich fish 2 or more days a week (defined as >0.5 g DHA or EPA/serving)
* Has a history of atrial fibrillation.
* Has been diagnosed with a significant psychiatric condition that might compromise adherence to study protocols, including eating disorders, schizophrenia, bipolar (manic phase), severe personality disorders, severe major depressive, severe anxiety disorders, and substance use disorders.
* Have an allergy to the study oils.
* Have received other investigational agents within the past 6 months.
* Currently on a weight reducing diet or has lost >5% body weight in the past 6 months.
* Currently using GLP-1
* Currently using prescribed anticoagulants or have a blood clotting problem or disease that causes excessive bleeding or been told by a physician that you have an increased risk of serious bleeding
* Currently using oral steroids
* Perceivably unable or unwilling to use acetaminophen in place of aspirin (including low dose regimen), NSAIDS, or other COX-2 inhibitors.
* Perceivably unable or unwilling to refrain from using anti- inflammatory supplements (including n-3 supplements).
* Perceivably unable or unwilling to refrain from using montelukast-type of allergy medications.
* Run-in failure

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean change in circulating arachidonic acid (ARA) between baseline and the end of each 12-week treatment period | From enrollment to end of phase 2 treatment (week 36)
  This outcome evaluates the within-subject change in circulating arachidonic acid. Measurements are collected at baseline and at the end of each 12-week treatment phase in a 36-week randomized, double-blind, placebo-controlled crossover trial.
Mean change in the ARA:DGLA ratio between baseline and the end of each 12-week treatment period | From enrollment to the end of Phase II intervention at 32 weeks.
  This outcome assesses the within-subject change in the ratio of arachidonic acid (ARA) to dihomo-γ-linolenic acid (DGLA), calculated using molar concentrations, from baseline to the end of each 12-week treatment period. A higher ARA:DGLA ratio reflects greater FADS1 enzymatic activity. Ratios are calculated using plasma phospholipid fatty acid levels measured by mass spectrometry in a 36-week randomized, double-blind, placebo-controlled crossover trial.
Mean change in the ARA:EPA ratio between baseline and the end of each 12-week treatment period. | From enrollment to the end of treatment Phase II at 32 weeks.
  This outcome assesses the within-subject change in the ratio of arachidonic acid (ARA) to eicosapentaenoic acid (EPA), calculated using molar concentrations, from baseline to the end of each 12-week treatment period. A lower ARA:EPA ratio indicates a shift toward greater omega-3 fatty acid abundance. Ratios are derived from plasma phospholipid fatty acid levels measured by mass spectrometry in a 36-week randomized, double-blind, placebo-controlled crossover trial.
Genotype-dependent differences in the effect of omega-3 supplementation on circulating arachidonic acid (ARA) levels. | From enrollment to end of phase 2 treatment (week 36)
  This outcome assesses whether the magnitude of change in circulating arachidonic acid (ARA), measured in micrograms per milliliter (µg/mL) of plasma phospholipids, differs by FADS genotype. The analysis compares within-subject treatment effects (omega-3 supplementation vs placebo) across genotype groups (e.g., GG, GT, TT) to evaluate genotype-dependent modification of response. ARA is measured at baseline and at the end of each 12-week treatment period in a 36-week randomized, double-blind, placebo-controlled crossover trial. Genotyping is performed using validated single nucleotide polymorphism (SNP) assays.
Genotype-dependent differences in the effect of omega-3 supplementation on the ARA:DGLA ratio | From enrollment to end of Phase II treatment (Week 36)
  This outcome assesses whether the magnitude of change in the ratio of arachidonic acid (ARA) to dihomo-γ-linolenic acid (DGLA), calculated using molar concentrations, differs by FADS genotype. The analysis compares within-subject treatment effects across genotype groups (e.g., GG, GT, TT) to evaluate genotype-dependent modification of response. ARA:DGLA ratio is derived from plasma phospholipid fatty acid levels measured at baseline and at the end of each 12-week treatment period in a 36-week randomized, double-blind, placebo-controlled crossover trial. Genotyping is conducted using validated SNP assays.
Genotype-dependent differences in the effect of omega-3 supplementation on the ARA:EPA ratio | From enrollment to end of Phase II treatment (Week 36)
  This outcome assesses whether the magnitude of change in the ratio of arachidonic acid (ARA) to eicosapentaenoic acid (EPA), calculated using molar concentrations, differs by FADS genotype. The analysis compares within-subject treatment effects across genotype groups (e.g., GG, GT, TT) to evaluate genotype-dependent modification of response. The ARA:EPA ratio is calculated from plasma phospholipid fatty acid levels measured at baseline and at the end of each 12-week treatment period in a 36-week randomized, double-blind, placebo-controlled crossover trial. Genotyping is performed using validated SNP assays.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Arizona Cancer Center, Tucson, Arizona
  - Georgetown University, Washington D.C., District of Columbia

IPD SHARING:
Plan to Share IPD: Undecided